CLINICAL TRIAL: NCT01750515
Title: Acupuncture as an Adjunctive Treatment for Hepatitis C Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assy Nimer (Other Government)
Responsible Party: Sponsor-Investigator, Assy Nimer, Prof. Assy Nimer, Ziv Hospital
Organization: Ziv Hospital (Other Government)
Other Study IDs: 0094-12-ZIV
Record Dates: First submitted 2012-11-26; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Hepatitis C (HCV); Acupuncture
Keywords: Acupuncture; Hepatitis C (HCV)
MeSH Terms: conditions — Hepatitis C | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group - acupuncture treatment (Experimental)
  Interventions: Device: Acupuncture
- Control group (No Intervention)

INTERVENTIONS:
Device: Acupuncture
  Arms: Intervention group - acupuncture treatment

SUMMARY:
Objective: to study the effect of Acupuncture on liver cirrhosis, SVR and health related quality of life in HCV patients receiving standard treatment (Peg Interferon+ Ribavirin).

Methods: 60 HCV patients receiving standard treatment (Peg Interferon+ Ribavirin) will undergo Serologic screening for hepatitis C virus (Anti-HCV EIAs and/or recombinant immunoblot assay) plus Transient Ultrasound Elastography (FibroScan) to achieve baseline characteristics(17,18,19). Patients will be randomized into intervention and control groups, 30 patients each.In the Intervention group each patient will receive an acupuncture treatment once a week for 12 consecutive weeks(Max 12, Min 8 treatments). Treatment protocol will be individualized for each patient according to TCM diagnosis. This treatment protocol is acceptable and has been published(20,21,22).In the control group patients will receive standard treatment alone, with no other intervention.

Data collection: after 12 weeks patients will again undergo Serologic screening for hepatitis C virus (Anti-HCV EIAs and/or recombinant immunoblot assay) plus Transient Ultrasound Elastography (FibroScan) in order to detect changes from baseline and group differences.

Inclusion criteria: adult patients with a confirmed HCV infection

Exclusion criteria:

Under 18 years Can not receive standard Peg interferon+ ribavirin treatment for any reason Psychiatric diagnosis Anaemia of hematologic origin Diabetic patient with uncontrolled diabetes Congestive heart failure, arrhythmia Hepatocellular carcinoma HIV infection Hepatitis B infection Auto immune liver disease or alcoholic liver disease Study duration: 1 year Study Location: "Ziv" medical center, division of liver disease, Israel

DETAILED DESCRIPTION:
Background:

Hepatitis C is an infectious disease affecting primarily the liver, caused by the hepatitis C virus (HCV). HCV is a worldwide problem, An estimated 130-170 million people worldwide are infected with HCV, in Israel there are an estimated 80,000 patients. Most patients infected with HCV have chronic liver disease, which can progress to cirrhosis and Hepatocellular carcinoma (HCC). Chronic infection with HCV is one of the most important causes of chronic liver disease and the most common indication for orthotropic liver transplantation (OLT) in the United States. Medical care costs associated with the treatment of HCV infection in the United States are estimated to be more than $600 million a year.

Chronic hepatitis C infection and chronic active hepatitis are slowly progressive diseases and result in severe morbidity in 20-30% of infected persons. Although acute HCV infection is usually mild, chronic hepatitis results in at least 75% of patients. Cirrhosis develops in 20-50% of patients with chronic hepatitis C infection. Liver failure and Hepatocellular carcinoma can eventually result. Hepatocellular carcinoma occurs in 11-19% of patients . The diagnosis of acute or chronic HCV infection generally requires testing of serum for both antibody to HCV (anti-HCV) and for HCV RNA. The recombinant immunoblot assay is used to confirm HCV infection. A sensitive quantitative HCV RNA assay is recommended for diagnosis because it also provides information on the level of virus which is helpful in management of the disease.

Combination therapy with pegylated interferon Alfa (PEG-IFN Alfa) and the nucleoside analogue ribavirin is the current standard of care in patients infected with HCV. Treatment of chronic HCV infection has 2 goals. The first is to achieve sustained eradication of HCV (ie, sustained virologic response [SVR]), which is defined as the persistent absence of HCV RNA in serum 6 months or more after completing antiviral treatment. The second goal is to prevent progression to cirrhosis, Hepatocellular carcinoma (HCC), and decompensated liver disease requiring liver transplantation.

Adverse effects are common with IFN and ribavirin combination therapy. Approximately 75% of patients experience one or more of adverse effects. Common adverse effects are :

1. Flulike symptoms
2. Hematologic complications (ie, neutropenia, thrombocytopenia)
3. Depression
4. Low grade fever,
5. Nausea, loss of weight
6. Neuropsychiatric complications (ie, memory and concentration disturbances, visual disturbances, headaches, irritability)
7. Metabolic complications (gout). Adverse events are a major reason that patients decline or stop therapy altogether. Currently there are limited options of managing these side effects, while being especially problematic are the flu like symptoms and depression . Traditional Chinese medicine(TCM) has been found as an effective treatment for improving quality of life in various medical conditions including hepatitis. TCM also positively affects chronic inflammation and improves inflammation markers in chronic inflammatory diseases such as asthma, crohn's disease, sinusitis and chronic pelvic inflammation .

Acupuncture's effect on liver cirrhosis, SVR(sustained Viral Response) and health related quality of life in chronic HCV patients has yet to be studied.

Study Aim: to study the effect of acupuncture as an adjunctive treatment for chronic HCV patients receiving standard treatment (Peg Interferon+ Ribavirin).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a confirmed HCV infection

Exclusion Criteria:

* Under 18 years
* Can not receive standard Peg interferon+ ribavirin treatment for any reason
* Psychiatric diagnosis
* Anaemia of hematologic origin
* Diabetic patient with uncontrolled diabetes
* Congestive heart failure, arrhythmia
* Hepatocellular carcinoma
* HIV infection
* Hepatitis B infection
* Auto immune liver disease or alcoholic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel